CLINICAL TRIAL: NCT00199407
Title: A 12-week, Double Blind, Placebo-controlled, Randomized, Parallel Group, Multicenter, Fixed Dose Study to Evaluate the Efficacy and Safety of a 20 mg/d Oral Dose of KW-6002 (Istradefylline) as Treatment for Parkinson's Disease in Patients With Motor Response Complications on Levodopa/Carbidopa Therapy.
Brief Title: A Study of Istradefylline (KW-6002) for the Treatment of Parkinson's Disease in Patients Taking Levodopa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6002-US-013
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; levodopa; end of dose wearing off; OFF time
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Istradefylline (KW-6002)

SUMMARY:
To establish the efficacy of a 20 mg/day dose of istradefylline for reducing the percentage of OFF time in patients with advanced Parkinson's disease (PD) treated with levodopa.

DETAILED DESCRIPTION:
To establish the efficacy of a 20 mg/d dose of istradefylline for reducing the percentage of OFF time in patients with advanced Parkinson's disease (PD) treated with levodopa. Patients who meet entry criteria will be randomized in a 1 to 1 ratio to either istradefylline or matching placebo. Patients will be treated for 12 weeks and will have interim visits and end of treatment visit to assess the efficacy and safety of istradefylline as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. UK Parkinson's Disease Society (UKPDS) brain bank criteria (Step 1 and 2) for PD.
2. PD stages 2-4 in the OFF state for Modified Hoehn and Yahr Scale.
3. On levodopa/carbidopa for at least one year, stable dose in past 4 weeks.
4. Currently take at least three doses of levodopa/carbidopa per day.
5. Predictable end of dose wearing off.
6. Able to satisfactorily complete Hauser version of a Parkinson's diary.
7. Have an average of 180 minutes of OFF time on two 24 hour diaries.
8. Be at least 30 years of age.

Exclusion Criteria:

1. Neurosurgical treatment for PD.
2. History of psychosis.
3. Diagnosis of atypical parkinsonism, secondary parkinsonism variant or Parkinson's plus syndromes.
4. Diagnosis of cancer within 5 years.
5. Mini-mental status examination score of 25 or less.
6. History of seizures or neurologic malignant_syndrome.
7. Clinical depression.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230
Dates: Start 2004-06; Primary Completion 2005-11 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To establish the efficacy of a 20 mg/d dose of istradefylline for reducing the percentage of OFF time in patients with advanced Parkinson's disease (PD) treated with levodopa/carbidopa.

SECONDARY OUTCOMES:
To evaluate the efficacy of a 20 mg/d dose of istradefylline for reducing the total hours of OFF time.
To evaluate the change in percentage of ON time (without dyskinesia, with dyskinesia, with non-troublesome dyskinesia, and with troublesome dyskinesia).
To evaluate the change in Unified Parkinson's Disease Rating Scale (UPDRS) Motor Examination score (part III) and/or in Activities of Daily Living (ADL) score (part II).
To evaluate the change in Parkinson's Disease Questionnaire (PDQ-39) and Medical Outcomes Study 36-item Short Form (SF-36).
To evaluate the change in the Patient Global Impression - Improvement scale (PGI-I).
To evaluate change in the Clinical Global Impression - Severity of Illness scale (CGI-S).
To evaluate the safety of a 20 mg/d dose of istradefylline.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sussman, MD, Study Director — Kyowa Kirin, Inc.
Locations (1):
- Kyowa Pharmaceutical Inc., Princeton, New Jersey, United States